CLINICAL TRIAL: NCT02390089
Title: Airway Protection Deficits According to Stimulus Type in Parkinson's Disease
Brief Title: Cough According to Stimulus Type in PD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB201401059-N; 1R21DC014567-01 (NIH)
Record Dates: First submitted 2015-02-19; First posted 2015-03-17 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Parkinson's Disease
Keywords: Dysphagia; Cough; Aspiration pneumonia
MeSH Terms: conditions — Parkinson Disease; Deglutition Disorders; Cough; Pneumonia, Aspiration | interventions — Weather; Nebulizers and Vaporizers

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Healthy control (Active Comparator): Healthy age-matched adult participants with no history of Parkinson's disease Participants in this group will receive capsaicin vapor cough provocation test. The vapor will be delivered using a small hand-held nebulizer.
  Interventions: Drug: Capsaicin vapor; Device: Nebulizer
- Parkinson's disease - no PA (Experimental): People with Parkinson's disease without penetration or aspiration during swallowing; based on results of videofluoroscopic swallow evaluation. Participants in this group will receive capsaicin vapor and fog cough provocation test using a small, hand-held nebulizer.Participants in the group will also receive a fluoroscopic swallow evaluation.
  Interventions: Drug: Capsaicin vapor; Other: fog; Radiation: Videofluoroscopic swallow evaluation; Device: Nebulizer
- Parkinson's disease - PA (Experimental): People with Parkinson's disease with penetration or aspiration during swallowing;based on results of videofluoroscopic swallow evaluation.Participants in this group will receive capsaicin vapor and fog cough provocation test using a small, hand-held nebulizer. Participants in the group will also receive a fluoroscopic swallow evaluation.
  Interventions: Drug: Capsaicin vapor; Other: fog; Radiation: Videofluoroscopic swallow evaluation; Device: Nebulizer

INTERVENTIONS:
Drug: Capsaicin vapor — Single-breath and continuous inhalation paradigm to induce cough.
  Other Names: hot pepper vapor
Other: fog — Continuous inhalation of fog until a cough is produced, or up to 60 seconds (whichever is shortest)
  Other Names: aerosolized water
  Arms: Parkinson's disease - PA; Parkinson's disease - no PA
Radiation: Videofluoroscopic swallow evaluation — Fluoroscopic evaluation of oropharyngeal swallowing function.
  Other Names: Swallow study; Modified barium swallow study
  Arms: Parkinson's disease - PA; Parkinson's disease - no PA
Device: Nebulizer — A hand-held nebulizer will be used to aerosolize the capsaicin and water solutions. Participants will inhale through the device's mouthpiece, and cough if they need to.

SUMMARY:
Aspiration pneumonia (APn) occurs at a higher rate in patients with Parkinson's disease (PD) versus healthy adults. This is of particular public health concern given that death secondary to aspiration pneumonia and lung infection is a leading cause of death in persons with PD. Swallowing and cough function are affected in PD, putting people with PD at significant risk for uncompensated aspiration (aspiration without adequate cough response). One challenge in the management of airway protective deficits related to PD is the chronic and progressive nature of the disease, where swallowing dysfunction appears subtly in the form of microaspiration, reducing the perceived urgency of the swallowing disorder by both clinicians and patients. The long-term goal of this research is to advance the management of airway protection deficits in patients with neurodegenerative disease in order to decrease morbidity and mortality due to aspiration related lung infection. The objective here is to further specify deficits leading to uncompensated airway compromise in PD in order to advance the clinical management of these patients, leading to an immediate positive impact.

DETAILED DESCRIPTION:
The study will be completed in one visit, and take about an hour. All study procedures are done in the investigators quiet clinical research area at the Center for Movement Disorders and Neurorestoration (Room 7). If participants agree to be in this research study, after participants sign the informed consent form, the investigators will ask participants some questions related to participants health history. These questions include:

Do participants have a history of any breathing disorders or diseases (asthma, emphysema/chronic obstructive pulmonary disease (COPD), etc), or severe chest injury?

* Do participants have any history of stroke, or any neurologic disease besides Parkinson's disease?
* Have participants smoked in the last 5 years?
* Have participants had any chest infections within the last 5 the weeks?
* Do participants have a history of head and neck cancer?
* Are participants allergic to capsaicin, hot peppers, Zostrix cream, or other medicines?

The investigators will ask these questions to make sure participants do not have a history of any illnesses that would affect their ability to cough or that would make it unsafe for them to participate. If participants answer yes to any of these questions, they will not be able to continue in the study.

Next, the investigators will begin to measure participants reflex cough. First, the investigators will attach a small microphone with a clip to participants shirt that will record participants cough responses. The investigators will have participants inhale a "hot pepper" vapor at five different concentrations. The hot pepper vapors will be separately delivered through a mouthpiece attached to a hand-held nebulizer (a device that makes vapors out of liquids). The investigators will deliver each type of vapor to participants 3 times each for a total of 15 presentations. After inhaling each vapor and coughing if participants need to, the investigators will ask participants to rate their urge to cough using a scale of 0-10, with 0 equaling no urge to cough, and 10 equaling the greatest urge to cough. If participants do not cough to any of the vapors, the investigators will present one final stronger dose. There will be a 2 minute break in between each presentation of the vapor, and water will be available at all times throughout the study. This will take approximately 40 minutes.

Next, the investigators will continue to measure participants reflex cough using a slightly different test. The investigators will have participants inhale water vapor (fog) and a low concentration of hot pepper vapor. Both types of vapor will be in separate nebulizers, like the ones the investigators just used. For these vapors, participants will breathe in and out through the nebulizer's mouthpiece until participants cough, or for up to 1 minute. The investigators will try each one 3 times, for a total of 6 tries.

ELIGIBILITY:
Inclusion Criteria:

* Within age limits
* For PD group: confirmed diagnosis of idiopathic parkinson's disease

Exclusion Criteria:

* Uncontrolled hypertension
* Difficulty complying due to neuropsychological dysfunction (i.e., severe depression)
* Allergy to capsaicin or hot peppers
* History of head or neck cancer
* Neurological disorders other than PD (i.e., stroke, etc.)

  1. control participants only: any history of neurologic disorders including PD
* History of smoking in the last 5 years
* Breathing disorders or diseases

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2015-04; Primary Completion 2017-02-10 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Urge-to-cough sensitivity | 30 minute
  Slope of the line created by plotting urge-to-cough (scale of 1-11) with capsaicin concentration (5 doses of increasing intensity).
Positive/negative cough response | 10 minutes
  A positive response is 2 coughs produced to 2/3 trials of the stimulus

SECONDARY OUTCOMES:
Latency | 10 minutes
  Time from stimulus presentation to cough produced.
Cough sensitivity threshold | 30 minutes
  the lowest concentration of capsaicin that elicits a perceived urge to cough of 1 (very slight) in at least 2/3 trials
Cough motor threshold | 30 minutes
  the lowest concentration of capsaicin that elicits at least 2 cough responses in 2/3 trials

OTHER OUTCOMES:
Swallowing group | 20 minutes
  The total number of participants with and without penetration or aspiration of material to the airway during swallow evaluation. Two groups will be identified, those with penetration or aspiration (PD-PA) and those without (PD).

CONTACTS AND LOCATIONS:
Overall Officials: Karen W Hegland, PHD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Center for Movement Disorders and Neurorestoration, Gainesville, Florida, United States